CLINICAL TRIAL: NCT02151084
Title: A Randomized Phase II Trial of MEK Inhibitor Selumetinib (AZD6244) Combined Continuously or Sequentially With Cisplatin/Gemcitabine (CIS/GEM) Versus CIS/GEM Alone in Patients With Advanced Biliary Cancer
Brief Title: A Study of Different Dosing Schedules of Selumetinib With Cisplatin/Gemcitabine (CIS/GEM) Versus CIS/GEM Alone in Biliary Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIL-MEK
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Biliary Tract Carcinoma; Gallbladder Carcinoma
Keywords: randomized; selumetinib; tablets; cisplatin; gemcitabine; non-resectable; recurrent; metstatic
MeSH Terms: conditions — Gallbladder Neoplasms; Recurrence | interventions — AZD 6244; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Continuous Dosing) (Experimental): Run-In: Selumetinib, orally, BID for 7 days (Day -7 to Day -1)
  On treatment: Selumetinib, orally, BID from Day 1-21 of every 28 day cycle. Cisplatin/gemcitabine, intravenously, on Days 1 and 8 of every 28 day cycle.
  Interventions: Drug: Selumetinib; Drug: Cisplatin; Drug: Gemcitabine
- Arm B (Sequential Dosing) (Experimental): Run-In: Selumetinib, orally, BID for 5 days (Day -7 to Day -3) with 2 days washout
  On treatment: Selumetinib, orally, BID from Day 1-5 and 8-19 of every 28 day cycle.
  Cisplatin/gemcitabine, intravenously, on Days 1 and 8 of every 28 day cycle.
  Interventions: Drug: Selumetinib; Drug: Cisplatin; Drug: Gemcitabine
- Arm C (Standard Care) (Experimental): Cisplatin/gemcitabine, intravenously, on Days 1 and 8 of every 28 day cycle.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Selumetinib
  Other Names: AZD6244
  Arms: Arm A (Continuous Dosing); Arm B (Sequential Dosing)
Drug: Cisplatin
  Other Names: Platinol
Drug: Gemcitabine
  Other Names: Gemzar

SUMMARY:
This is a phase II study (the second stage of testing a new drug or new drug combinations) to see how useful two different schedules of study drug selumetinib with cisplatin and gemcitabine are compared to cisplatin and gemticabine alone in patients with biliary cancer.

Selumetinib, an oral drug which plays an important role in the regulation of cell growth (MEK 1/2 inhibitor) has been shown to shrink tumours in patients with biliary cancer and other types of human cancers. Selumetinib has also been shown to shrink tumours when given in combination with cisplatin and gemcitabine in research studies done in animals and in some patients with biliary tract cancer. Cisplatin and gemcitabine are intravenous drugs that work by damaging DNA in tumor cells so that they are unable to grow and divide.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable, recurrent or metastatic, measurable biliary tract cancer or gall bladder cancer
* No prior systemic therapy
* Performance status 0, 1, or 2
* Age 18 years or older
* Estimated life expectancy > 3 months
* Adequate hematological, liver, renal function
* No evidence of active uncontrolled infection
* Capable of giving written consent
* Acceptable recovery of previous side effects

Exclusion Criteria:

* Progressing within 3 or 6 months of receiving certain treatments
* Prior chemotherapy for non-resectable or metastatic disease or a MEK inhibitor
* Progressing within 6 months of adjuvant treatment.
* May not have received prior chemotherapy for non-resectable/metastatic disease.
* Prior MEK, RAS, or RAF inhibitors or history of hypersensitivity to study drugs.
* Ampullary carcinoma
* Incomplete recovery from previous surgery
* Undergoing treatment with curative intent
* Prior malignancy that could interfere with the response evaluation
* Severe or uncontrolled systemic diseases or lab finding that makes it undesirable for patient to participate
* Any psychiatric or other disorder likely to impact consent
* Pregnant or breastfeeding
* Patients with significant cardiac-related issues
* History of eye-related issues.
* Systemic disease, active infection, bleeding diatheses or renal transplant, including hep B, hep C or HIV
* Receiving potent inhibitors or inducers of CYP3A4/5, CYP2C19 and CYP1A2 can continue with caution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in tumor size in millimetres | 10 weeks post initiation of therapy
  Response Evaluation Criteria in Solid Tumors (RECIST 1.1)

SECONDARY OUTCOMES:
Number of participants with objective response and/or stable disease | 6 months post initiation of therapy
Percentage of patients without progressive disease | 10 weeks post initiation of therapy
Progression-free survival in months | Enrollment to disease progression or death
Overall survival in months | Time from enrollment to date of death
Total incidence of adverse events | 2 years
Total rate of grade 3 and 4 toxicities | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Knox, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada